CLINICAL TRIAL: NCT04641234
Title: Belgian Retrospective Chart Review Evaluating Treat-and-extend With Eylea® in Treatment naïve Patients With Neovascular Age-related Macular Degeneration.
Brief Title: A Study Reviewing Medical Records to Learn More About Treat-and-extend With Eylea in Patients With Neovascular Age-related Macular Degeneration (nAMD).
Acronym: BELUGA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21573
Record Dates: First submitted 2020-11-20; First posted 2020-11-23 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Retinal disorders; aflibercept; treat-and-extend
MeSH Terms: conditions — Retinal Diseases | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Adult Belgian patients diagnosed with neovascular age-related macular degeneration (nAMD) with treatment-naïve study eye.
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — As prescribed by the treating physician

SUMMARY:
In people with neovascular age-related macular degeneration (nAMD), the body makes too much of a protein called vascular endothelial growth factor (VEGF). This causes too many blood vessels to grow in a part of the eye called the macula. These blood vessels can damage the macula, causing dark spots and blurriness in central vision.

The study drug, aflibercept, works by reducing VEGF levels in the eye.It has already been approved for patients to receive as a treatment for nAMD in a fixed 8-weekly or treat-and-extend dosing regimen after having received 3 monthly doses at the start of treatment. In this study, the researchers want to learn more about how often patients received aflibercept and how their vision changed.

The study will include patients with nAMD who had not received treatment to reduce VEGF levels in the eye before. These patients will have started treatment with aflibercept between January 2016 and November 2018. The study will include about 330 men and women who are at least 18 years old.

All of the patients had received aflibercept eye injections based on their doctor's instructions. The researchers will use the patients' medical records from January 2016 to November 2020 to measure the following:

* the number of aflibercept eye injections the patients received
* how long the patients could wait between treatments
* the change in the patients' vision
* how many patients stopped treatment and why.
* associations between patient and disease characteristics at the start of treatment with the number of aflibercept injections and patient's vision during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) patients diagnosed with nAMD
* Anti-VEGF treatment-naïve
* Started Intravitreal (IVT) aflibercept treatment between 01 January 2016 and 30 November 2018
* Aflibercept treatment according to Treat-and-Extend (T&E) immediately after the loading dose
* Availability of medical records of aflibercept treatment.

Exclusion Criteria:

* Participation in an investigational program with interventions outside of routine clinical practice during the aflibercept treatment
* Patients with eye diseases that required surgery during the first 24 months of aflibercept treatment, e.g. advanced glaucoma, visually significant cataracts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients to be enrolled into the study must have been diagnosed with neovascular age-related macular degeneration (nAMD) and started anti-VEGF treatment with aflibercept.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Number of injections in the first 24 months of treatment | Retrospective analysis in the first 24 months of treatment (1 January 2016 - 30 November 2020)
Last injection interval in the 2nd year of treatment | Retrospective analysis in the first 24 months of treatment (1 January 2016 - 30 November 2020)

SECONDARY OUTCOMES:
Number of aflibercept injections during the 1st, 3rd and 4th year of treatment | Retrospective analysis from 01-Jan-2016 to 30-Nov-2020
Last injection interval in the 1st, 3rd and 4th year | Retrospective analysis from 01-Jan-2016 to 30-Nov-2020
Most stable interval between aflibercept injections in the 2nd, 3rd and 4th year | Retrospective analysis from 01-Jan-2016 to 30-Nov-2020
  Definition of 'most stable injection interval according to the ophthalmologist
Number of monitoring visits during each year of the study | Retrospective analysis from 01-Jan-2016 to 30-Nov-2020
Change in best corrected visual acuity (BCVA) from baseline to 90 days and after each year in the study | Retrospective analysis from 01-Jan-2016 to 30-Nov-2020
  BCVA is assessed by ETDRS (Early Treatment Diabetic Retinopathy Study) or Snellen chart with conversion to ETDRS.
Central retinal thickness (in μm) measured by Optical coherence tomography (OCT) | Retrospective analysis from 01-Jan-2016 to 30-Nov-2020
  Retinal and lesion characteristics were evaluated using spectral domain optical coherence tomography (OCT).
Number of patients with presence of fluid or anatomical parameters (IRF/SRF/PED) | Retrospective analysis from 01-Jan-2016 to 30-Nov-2020
  IRF:Intra-Retinal Fluid/ SRF: Sub-Retinal Fluid / PED:Pigment Epithelial Detachment
Number of patients with absence of fluid or anatomical parameters (IRF/SRF/PED) | Retrospective analysis from 01-Jan-2016 to 30-Nov-2020
Reason for discontinuation of aflibercept treatment after 24 months | Retrospective analysis from 01-Jan-2016 to 30-Nov-2020
  Reasons : Adverse event, lack of efficacy, remission and stop monitoring, remission and start monitor-and-extend, reimbursement issues, patients' decision, unknown
Number of patients discontinuing aflibercept treatment within the first 24 months | Retrospective analysis from 01-Jan-2016 to 30-Nov-2020
Reason for discontinuation of aflibercept treatment during first 24 months | Retrospective analysis from 01-Jan-2016 to 30-Nov-2020
  Reasons :Adverse event, lack of efficacy, remission and stop monitoring, remission and start monitor-and-extend, reimbursement issues, patients' decision, unknown
Number of patients discontinuing aflibercept treatment after 24 months | Retrospective analysis from 01-Jan-2016 to 30-Nov-2020

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.